CLINICAL TRIAL: NCT02149017
Title: Phase 1 and Phase 2 Clinical Trials for the Evaluation of Pharmacokinetics, Safety, and Efficacy of SNUBH-NM-333(18F) in Alzheimer's Disease Patients and Healthy Volunteers.
Brief Title: Phase 1 and Phase 2 Clinical Trials of SNUBH-NM-333(18F)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: SNUH-NM-333 ligand effect was judged to be insufficient.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jong Inn Woo, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUBH-NM-333(18F)
Record Dates: First submitted 2014-05-19; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Alzheimer Disease
Keywords: amyloid plaque; Positron-Emission Tomography; radiopharmaceuticals
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SNUBH-NM-333(18F), Safety, Efficacy (Experimental): 10 young controls, 10 cognitively normal elderly, and 10 Alzheimer's disease patients
  Interventions: Radiation: SNUBH-NM-333(18F)

INTERVENTIONS:
Radiation: SNUBH-NM-333(18F) — 5-10 mCi

SUMMARY:
To evaluate pharmacokinetics, safety and efficacy of SNUBH-NM-333(18F), a new diagnostic radiopharmaceutical for PET imaging of amyloid plaques, in Alzheimer's disease patients and healthy volunteers.

DETAILED DESCRIPTION:
The investigators will perform whole-body and brain kinetic modeling of SNUBH-NM-333(18F) and optimize the image acquisition procedure.

Five young healthy subjects will be participated in Whole-body positron emission tomography /computed tomographic (PET/CT) scans from the midfemoral position to the head after approximately 5-10 mCi of SNUBH-NM-333(18F) injection. For brain PET/CT amyloid imaging, another five young healthy subjects will be scanned dynamically during windows of 0-180 min after injection of SNUBH-NM-333(18F), with arterial sampling.

The investigators will compare different analysis methods of compartmental modeling and standardized uptake value ratios and determine the optimal acquisition window. And then 10 AD patients and 10 elderly healthy controls will also be participated in brain amyloid imaging to compare SNUBH-NM-333(18F) brain retention in AD patients versus healthy elderly.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young controls who are 20 - 30 years old and have no subjective memrory complaints
* Cognitively normal elderly who have Clinical Dementia Rating score of 0
* Alzheimer's disease (AD) patients who met both the DSM-IV criteria for dementia and NINCDS-ADRDA criteria for probable AD

Exclusion Criteria:

* any present serious medical, psychiatric, or neurological disorder that could affect mental function; evidence of focal brain lesions on MRI; the presence of severe behavioral or communication problems

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Distribution volume ratio (DVR) | Whole-body positron emission tomography /computed tomographic (PET/CT) scans will be performed within 30 days after screening.
  DVR = Distribution volume of region of interest/Distribution volume of reference region

SECONDARY OUTCOMES:
Standardized uptake value ratio (SUVr) | Whole-body positron emission tomography /computed tomographic (PET/CT) scans will be performed within 30 days after screening.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Eun Kim, MD, PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea